CLINICAL TRIAL: NCT05070039
Title: Value of Cortactin Expression in Invasive and Non-invasive Urinary Bladder Urothelial Carcinoma in Egyptian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, lecturer of pathology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Soh-Med-21-09-44
Record Dates: First submitted 2021-09-19; First posted 2021-10-06 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Urothelial Carcinoma
Keywords: Cortactin; Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: formalin fixed and paraffin embedded blocks of urinary bladder malignant neoplasms will be obtained and sectioned. from each block, one tissue section will be stained by H&E, other section will be stained immunohistochemically by anti Cortactin antibodies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with invasive and non invasive urothelial carcinoma (Other): patients with urothelial carcinoma will be subjected to radical cystectomy or trans uretheral resection of the tumor, specimens will be sent to the pathology lab. to be examined.
  Interventions: Genetic: Expression of Cortactin anti body

INTERVENTIONS:
Genetic: Expression of Cortactin anti body — assessment of Cortactin immunohistochemical expression in invasive and non-invasive urothelial carcinoma.

SUMMARY:
Urothelial carcinoma is the ninth most common malignant neoplasm worldwide. nearly in all human tumors, actin filaments are involved in lamellopodia or cellular extensions. Cortactin is involved in fixing the actin assembly to enhance cellular penetration. Assessment of Cortactin expression in invasive and non-invasive urothelial carcinoma and recording any significant different expressions may have benefits in developing more effective anticancer chemotherapeutic agents.

DETAILED DESCRIPTION:
Bladder carcinoma is the 9th most prevalent cancer worldwide. Mostcases are diagnosed in men. Bladder carcinoma is categorized into three disticly different categories; non- muscle invasive, muscle invasive and metastatic bladder carcinoma. Vast majority of all bladder carcinomas are diagnosed as urothelial carcinoma (UC). Squamous cell carcinoma (SCC), adenocarcinoma and other rare types represent the remaining 10%. In Egypt, bladder carcinoma is ranked as the most prevalent cancer . The most important etiological causes for such disease in Egypt are festation by S. haematopium and Cigarette smoking. Cortactin is a 63-65 kDa protein, encoded by a gene located on 11q13. Cortactin activates and binds to Arp2/3 and stabilizes the branched Actin networks. Invadopodia are Actin-rich cellular protrusions, associated with enhanced proteolytic activities in the invasive regions of carcinomas. it is also incorporated in invadopodia, Cortactin expression is enhanced once or rapidly following secretions of transmembrane metalloproteinase, MT1-MMP. Extracellular matrix (ECM) proteolytic cleavage develops soon after secretion of MT1-MMP and Cortactin. increased secretion of Cortactin was studied in a lot of malignant tumors, including melanoma, mammary, pancreatic duct, hepatocellular and colorectal adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary urinary bladder carcinoma.

Exclusion Criteria:

* patients received chemotherapeutic agents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment and correlating Cortactin expression in invasive and non-invasive urothelial carcinoma. | 6 months
  immunohistochemical staining of tumor sections and correlating the immuno-expresion of Cortactin to different tumor parameters as tumor grade, stage and status of lymph nodes involved, inorder to detect the prognostic role of Cortactin in urothelial carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Maisa Hashem Mohammed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No